CLINICAL TRIAL: NCT06987825
Title: Chinese Atrial Fibrillation Registry
Acronym: China-AF
Status: Recruiting | Type: Observational
Sponsor: Beijing Anzhen Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: KS2025087
Record Dates: First submitted 2025-05-16; First posted 2025-05-23 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2025-05

CONDITIONS: Atrial Fibrillation (AF)
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This prospective, observational cohort study aims to establish a long-term registry of adult patients with atrial fibrillation (AF) in China to comprehensively characterize patient profiles and evaluate real-world management and outcomes over time. The objectives of the study are to:

* Describe the demographic, clinical, and treatment characteristics of AF patients across different stages of disease progression.
* Assess the effectiveness and safety of various AF treatment strategies, including oral anticoagulation, catheter ablation, and left atrial appendage closure, in routine clinical practice.
* Identify patient- and treatment-related factors that influence therapeutic outcomes.
* Explore the role of advanced technologies and artificial intelligence in improving procedural performance, risk stratification, and clinical decision-making in AF care.

Participants will undergo standardized baseline evaluation and longitudinal follow-up to collect data on heart rhythm monitoring, treatment exposures, healthcare utilization, clinical events, and patient-reported outcomes. This cohort will generate real-world evidence to inform personalized and evidence-based management of AF.

DETAILED DESCRIPTION:
This prospective, multicenter observational registry aims to collect standardized clinical data on adults with atrial fibrillation (AF) across over 30 hospitals in China. The study reflects real-world clinical practice and does not interfere with treatment decisions.

Baseline and follow-up data will be collected using standardized forms, including demographics, medical history, cardiovascular risk factors, laboratory and imaging results, medication use, and-when applicable-procedural details for catheter ablation, such as energy source and complications.

Follow-up will be conducted at 1, 2, 3, and 6 months after enrollment, and every 6 months thereafter. Data include ECG monitoring, medication updates, hospitalizations, adverse events (e.g., stroke, bleeding, cardiovascular death), and healthcare utilization. Quality of life, cognitive, and psychological assessments may also be collected.

All treatments are determined by physicians as part of usual care. The registry provides internal feedback on potential treatment issues and generates periodic, anonymized summaries for participating centers.

The study aims to inform clinical practice and support real-world evidence generation to improve AF management in China.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years;
2. Documented atrial fibrillation episode lasting >30 seconds confirmed by electrocardiogram (ECG), Holter monitor, implantable cardiac monitor, or wearable ECG device
3. Signed informed consent and willingness to participate in follow-up

Exclusion Criteria:

1. Atrial fibrillation due to a reversible cause (e.g., transient secondary AF)
2. Presence of comorbid conditions associated with an expected life expectancy of less than 1 year

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults (≥18 years) with documented atrial fibrillation enrolled from multiple hospitals across China.
Sampling Method: Non-Probability Sample
Enrollment: 100000 (Estimated)
Dates: Start 2011-08-01 (Actual); Primary Completion 2035-12-31 (Estimated); Study Completion 2035-12-31 (Estimated)

PRIMARY OUTCOMES:
All-cause death | 10 years
  Death due to any cause.

SECONDARY OUTCOMES:
Ischemic Stroke | 5 years
  An acute episode of neurological dysfunction caused by focal cerebral, spinal, or retinal infarction, confirmed by neuroimaging (CT or MRI) or clinical criteria consistent with permanent tissue injury.
Hemorrhagic Stroke | 5 years
  Bleeding within the brain parenchyma or into the subarachnoid space due to rupture of cerebral blood vessels. Subtypes include intracerebral hemorrhage and subarachnoid hemorrhage.
Transient ischemic attack (TIA) | 5 years
  A sudden onset of neurological deficit lasting less than 24 hours.
Cardiovascular Death | 5 years
  Death resulting from cardiovascular causes, including acute myocardial infarction, sudden cardiac death, heart failure, stroke, fatal bleeding, or complications related to cardiovascular interventions.
Cardiovascular Hospitalization | 5 years
  Unplanned hospital admission primarily due to cardiovascular causes, including acute coronary syndrome, heart failure exacerbation, arrhythmia, stroke, cardiovascular procedures, or thromboembolic or bleeding complications.
Systemic Embolism | 5 years
  An acute arterial occlusion outside the central nervous system, confirmed by imaging or surgery, with clinical evidence of embolic origin. Events limited to pulmonary embolism are excluded.
Thromboembolic Death | 5 years
  Death that occurs in the context of a confirmed or suspected thromboembolic event, such as ischemic stroke or systemic embolism, without an alternative non-cardiovascular cause.
Major Bleeding | 5 years
  Defined according to the International Society on Thrombosis and Haemostasis (ISTH) as any of the following:
  (1)Fatal bleeding; (2) Symptomatic bleeding in a critical area or organ (e.g., intracranial, intraspinal, intraocular, pericardial, retroperitoneal); (3) A fall in hemoglobin of ≥2 g/dL (20 g/L), or leading to transfusion of ≥2 units of whole blood or red cells.
Clinically Relevant Non-Major Bleeding (CRNMB) | 5 years
  Any bleeding that does not meet the criteria for major bleeding but is associated with medical intervention, unscheduled physician contact, temporary interruption of treatment, or discomfort sufficient to interfere with daily activities.

CONTACTS AND LOCATIONS:
Overall Officials: Changsheng Ma, MD, Principal Investigator — Beijing Anzhen Hospital
Locations (2):
- China (2):
  - Beijing Anzhen Hospital, Beijing, Beijing Municipality
  - Sir Run Run Shaw Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang